CLINICAL TRIAL: NCT00129948
Title: An Open-Label, Single-Arm, Multi-Center, Phase II Study of Troxatyl™ (Troxacitabine) Administered by Continuous Infusion in Patients With Acute Myeloid Leukemia (AML) in Second Salvage
Brief Title: Study for Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SGX Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD758-216; NCT00310193 (obsolete NCT alias)
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute myeloid leukemia; AML; refractory; relapsed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — troxacitabine

INTERVENTIONS:
Drug: Troxatyl™ (troxacitabine)

SUMMARY:
This is a phase 2, single-arm, open-label, multi-center study to establish the safety and efficacy of Troxatyl™ (troxacitabine) administered as a continuous infusion for 5 days to subjects with AML.

DETAILED DESCRIPTION:
This is a phase 2, single-arm, open-label, multi-center study to establish the safety and efficacy of Troxatyl™ (troxacitabine) administered as a continuous infusion for 5 days to subjects with AML. The study will primarily assess the complete response (CR) rate of a 5-day continuous infusion of troxacitabine at 12 mg/m2/day given as second salvage therapy in adult patients with AML, with secondary objectives to determine the overall, relapse-free and event-free survival and remission duration; to determine the duration of response; to determine the complete response with incomplete platelet recovery (CRp) rate; to evaluate the tolerability and safety of 5-day continuous intravenous (IV) infusion of troxacitabine; and to determine the relationship between troxacitabine plasma concentrations, anti-leukemic activity and adverse events. Additional cycles of treatment may be given at the investigator's discretion, provided that the subject does not have progressive disease or experience a dose limiting toxicity. Bone marrow transplantation in responding subjects will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute myeloid leukemia (AML) in the second salvage setting: refractory to two prior courses of therapy or primary refractory without response to two previous courses of leukemia therapy.
* Patients must have received at least two previous courses of induction chemotherapy to be considered in the second salvage setting.
* Patients who are in second relapse, must have had a duration of their second CR or CRp of less than six months.
* Subjects must have adequate organ and immune function as indicated by the following laboratory values:

  * Creatinine clearance ≥ 45 mL/min and ≤ 125 mL/min;
  * Total bilirubin ≤ 2.0 mg/dL (≤ 34.2 µmol/L);
  * AST (SGOT) and ALT (SGPT) ≤ 3 x upper limit of normal (ULN).
  * Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of < 2, and an estimated life expectancy of at least eight weeks.

Exclusion Criteria:

* Clinical evidence of active central nervous system (CNS) leukemic involvement
* Active and uncontrolled infection
* Uncontrolled medical problems unrelated to the malignancy that impair patient ability to give informed consent or unacceptably reduce the safety of the proposed treatment
* Neurologic or psychiatric disorders that would interfere with informed consent or study follow-up
* Known or suspected intolerance or hypersensitivity to Troxatyl® or closely related compounds such as lamivudine or any of the stated ingredients
* A recent history of alcohol or other substance abuse
* Subjects who have used another investigational agent or participated in a clinical trial within the last 14 days prior to enrolment
* Females with a positive pregnancy test at screening
* Subjects who have previously been enrolled into this study and subsequently withdrew

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211
Dates: Start 2005-07; Study Completion 2007-10

PRIMARY OUTCOMES:
To determine complete response (CR) rate

SECONDARY OUTCOMES:
To determine the complete response with incomplete platelet recovery (CRp) rate, and recurrent disease (RD) rates
Efficacy and safety, preliminary evidence of the anti-tumor activity, determination of Troxatyl™ infusion pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giles, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (20):
- United States (20):
  - Scripps Clinic, La Jolla, California
  - USC-Norris Neuro-Oncology Program, Los Angeles, California
  - UCSD Moores Cancer Center, San Diego, California
  - Univ. of Florida, Baptist Cancer Center, Jacksonville, Florida
  - Winship Cancer Institute, Emory University Hosp., Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Harper Hospital - Karmanos Cancer Center, Detroit, Michigan
  - Univ. of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Cornell Campus, New York, New York
  - Wake Forest Univ. School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Univ. of South Carolina, Hematology/Oncology Division, Charleston, South Carolina
  - Univ. of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Morgantown Internal Medicine Group, Morgantown, West Virginia